CLINICAL TRIAL: NCT01836302
Title: Septic Shock and Delirium Because of rSO2 Abnormalities in Intensive Care Unit Patients (The SAD BRAIN Study)
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Duane Funk, Assistant Professor, University of Manitoba
Other Study IDs: B2011:138
Record Dates: First submitted 2013-04-16; First posted 2013-04-19 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Septic Shock; Delirium; Renal Failure
MeSH Terms: conditions — Shock, Septic; Delirium; Renal Insufficiency | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Cerebral Desaturation: We will compare the primary and secondary outcomes between the patients who experience cerebral desaturations and those that do not.
  Interventions: Other: Observation
- Patients without cerebral desaturation: We will compare the primary and secondary outcomes between the patients who experience cerebral desaturations and those that do not.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
Delirium in the ICU is a prevalent problem occurring in up to 80% of ICU patients. A potential cause of delirium in ICU patients could be cerebral hypoxia. Septic shock is associated with high rates of delirium.

The aim of this pilot study is two fold. First, to determine the feasibility and potential challenges of measuring cerebral oxygenation in ICU patients with severe sepsis and septic shock. And second, to see if the incidence and magnitude of cerebral desaturations correlated with ICU acquired delirium as measured by the Confusion Assessment Method (CAM) scores.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* Diagnosis of septic shock
* Require mechanical ventilation and vasopressor therapy

Exclusion Criteria:

* Previous stroke
* Dementia
* Recent Craniotomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Intensive Care Unit with Septic Shock
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Delirium | 28 Days

SECONDARY OUTCOMES:
Death | 28 Days

OTHER OUTCOMES:
Renal Failure | 28 Days
  Defined using RIFLE Criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences Center, Winnipeg, Manitoba, Canada